CLINICAL TRIAL: NCT04304742
Title: Retrospective Study Comparing Radiologist Diagnostic Performance Versus Artificial Intelligence (AI) for Hip Fracture Suspicion in Elderly Patients
Brief Title: Radiologist Diagnostic Performance Versus Artificial Intelligence (AI)
Acronym: RAVIA
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0126
Record Dates: First submitted 2020-03-09; First posted 2020-03-11 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Painful Hip; Fonctional Impotence After Minor Trauma (Fall)
Keywords: Medical imaging diagnosis; Frature detection; Artificial intelligence; Femoral neck fracture; Hip; X-ray; Radiography
MeSH Terms: conditions — Femoral Neck Fractures | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Suspicion of hip fracture: Suspicion of hip fracture
  Interventions: Procedure: hip standard radiography/ CT scan/ MRI

INTERVENTIONS:
Procedure: hip standard radiography/ CT scan/ MRI — hip standard radiography/ CT scan/ MRI

SUMMARY:
In France, femoral neck fracture is mainly detected with interpretation of pelvis/hip X-ray imaging (French Health Authority recommandation).

However, up to 10% of fractures are not identified or misdiagnosed, especially in patients admitted to the emergency department.

Indeed, radiologists may be subject to excessive work, wich cause the risk of inaccurate on X-rays diagnosis.

The Artificial intelligence (AI) begins study the detection of fratures on medical imaging.

In this retropective study, this technology developed by GLEAMER company is tested to evaluate the detection rate of hip fracture and specifically femoral neck fracture, compared to the radiologist diagnostic, in eldery patients admitted in emergency department.

AI could optimize the diagnostic performance of radiologists (increase of confidence level) and improve the efficiency of suspected fractures sorting from emergency department.

ELIGIBILITY:
Inclusion criteria:

* Patients aged 60 and older
* Minor trauma
* Admitted in emergency department for painful hip/fonctional impotence after minor trauma
* Takes at least a hip radiography

Exclusion criteria:

* Painful before the minor trauma
* Important trauma

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 60 and older, admitted to emergency department for painful hip/fonctional impotence after minor trauma.
  Patients take at least a hip radiography
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Detection rate of femoral neck fracture | 1 day
  Detection rate of femoral neck fracture

SECONDARY OUTCOMES:
Detection rate of other hip fracture | 1 day
  Detection rate of other hip fracture

CONTACTS AND LOCATIONS:
Overall Officials: Catherine CYTEVAL, MD.PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC